CLINICAL TRIAL: NCT06832917
Title: A Prospective Multicenter, Two-arm Parallel, Open-label, Randomised Phase III Study to Explore the Efficacy and Safety of Cadonilimab Plus Chemotherapy After Short-course Radiotherapy in Locally Advanced Rectal Cancer
Brief Title: Short-course Radiation (SCRT) Followed by 6 Cycles of Cadonilimab Plus MFOLFOX6 As Neoadjuvant Therapy for Patients with Locally Advanced Rectal Cancer (LARC): a Multicenter, Two-arm Parallel, Open-label, Randomised Phase III Trial (NeoCaCRT-III)
Acronym: NeoCaCRT-III
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wan He (Other)
Responsible Party: Sponsor-Investigator, Wan He, Prof. He, Shenzhen People's Hospital
Organization: Shenzhen People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shenzhen CRC-005
Record Dates: First submitted 2025-02-13; First posted 2025-02-18 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Rectal Cancer
Keywords: Mismatch repair-proficient (pMMR) or microsatellite stability(MSS); Locally advanced rectal cancer (LARC); Short course radiation (SCRT)
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AK104 plus (Experimental): SCRT followed by AK104 plus chemotherapy
  Interventions: Drug: AK104 plus; Drug: Chemo only
- Chemo only (Other): SCRT followed by chemotherapy
  Interventions: Drug: Chemo only

INTERVENTIONS:
Drug: AK104 plus — SCRT followed by 6 cycles of cadonilimab (AK104) plus mFOLFOX6 as neoadjuvant therapy for patients
  Arms: AK104 plus
Drug: Chemo only — Short-course radiation (SCRT) followed by 6 cycles of mFOLFOX6 as neoadjuvant therapy for patients

SUMMARY:
The goal of this clinical trial is to learn if neoadjuvant short-course radiation (SCRT) followed by 6 cycles of cadonilimab plus mFOLFOX6 works to treat patients with locally advanced rectal cancer (LARC). It will also learn about the safety of the combined regimen. The main questions it aims to answer are:

Does the neoadjuvant SCRT plus dual immunotherapy and chemotherapy can improve pathological complete response(pCR) rate? What medical problems do participants have when receiving chemotherapy plus cadonilimab compared to chemotherapy only?

Participants will:

Receiving cadonilimab plus mFOLFOX6 or mFOLFOX6 every 2 weeks for 3 months Visit the clinic once every 2 weeks for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 yeas and ≤79 years. The gender is not limited. 2. Histopathology confirmed the diagnosis of rectal adenocarcinoma. 3. Patients with rectal cancer based on endoscopic ultrasound and / or pelvic MRI contrast + contrast, chest CT, head MRI or CT + contrast, or PET / CT, staging criteria per AJCC 8th edition cancer stage, cT 3-T4 / N + M0.

  4. At least 20 unstained sections of formalin-fixed paraffin-embedded tumor tissue sections, or fresh tumor tissue, can be provided for genomic and proteomic testing.

  5. The Eastern Cooperative Oncology Group Performance status (ECOG PS) 0- 1. 6. Adequate bone marrow and organ function meets the following criteria:
  1. Neutrophil count (ANC)≥1.5×l09/L
  2. Platelet (PLT) ≥80×109/L
  3. Hemoglobin (Hb) level ≥90 g/L
  4. Total bilirubin level≤1.5×ULN
  5. Alanine aminotransferase (ALT) level≤3×ULN
  6. Aspartate aminotransferase (AST) level ≤3×ULN
  7. International normalized value (INR) or prothrombin time (PT) or activated partial thromboplastin time (aPTT) ≤1.5×ULN
  8. Serum creatinine (Cr) level ≤1.5×ULN
  9. Creatinine clearance #50 ml/min (Calculated according to the Cockcroft-Gault formula)

     Exclusion Criteria:
* 1. Previous history of severe hypersensitivity to other monoclonal antibodies or any component of AK 104.

  2. Preoperative pathology was diagnosed as squamous cell carcinoma or neuroendocrine tumor 3. Within 5 years before enrollment for malignancies other than colorectal cancer with negligible risk of metastasis or death (e. g., expected 5-year OS> 90%) and expected radical results after treatment (e. g., adequately treated cervical carcinoma in situ, basal or squamous cell skin carcinoma, localized prostate carcinoma for curative intent, ductal carcinoma in situ surgically treated with curative intent).

  4. Previous treatment against the PD-1 receptor or its ligand PD-L1 or the cytotoxic T lymphocyte-associated protein-4 (CTLA-4) receptor.

  5. History of autoimmune diseases, including but not limited to myasthenia gravis, myoitis, autoimmune hepatitis, series, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis related to antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, vasculitis, or glomerulnephritis; patients with autoimmune-related hypothyroidism were eligible for stable-dose thyroid hormone replacement therapy; patients with type 1 diabetes under control after a stable insulin regimen were eligible to participate in this study; 6. Receiving systemic immune stimulation drugs (including but not limited to interferon or IL-2) within 4 weeks prior to enrollment or within 5 half-lives of the drug (whichever is shorter); 7. Received systemic corticosteroids (> 10 mg/d of prednisone equivalent) or other systemic immunosuppressive agents (including but not limited to prednisone, prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF agents [anti-TNF]) within 2 weeks prior to enrollment. Local, ocular, intra-articular, nasal, and inhaled corticosteroids are permittedt; 8. Patients requiring baseline and subsequent MRI tumor evaluation with previous allergic reactions to intravenous contrast agents may use preventive steroids.

  9. Allowing the use of inhaled corticosteroids for chronic obstructive pulmonary disease, corticosteroid hydrochloride (e. g., flurohydrocortisone) in patients with orthostatic hypotension, and low-dose corticosteroid maintenance for adrenal cortical insufficiency.

  10. Patients with previous allogeneic bone marrow transplantation or previous solid organ transplantation.

  11. Idiopathic pulmonary fibrosis, drug-induced pneumonia, mechanical pneumonia (i. e. bronchiolitis obliterans), history of idiopathic pneumonia or chest CT scan at screening showed evidence of active pneumonia.

  12. Any live vaccine (e. g., vaccine against infectious diseases, such as influenza vaccine, varicella vaccine, etc.) within 4 weeks (28 days) before enrollment.13 Active infections, including tuberculosis (clinical diagnosis including clinical history, physical examination and imaging findings, and TB tests performed per local medical practice), hepatitis B {known HBV surface antigen (HBsAg) positive and HBVDNA 1000 cps / ml}, hepatitis C or human immunodeficiency virus (HIV antibody positive).

  13. Patients with prior or cured HBV infection (defined as hepatitis B core antibody [anti-HBc] positive and HbsAg negative) were to be eligible to participate in the study only if HBVDNA was negative (HBVDNA˂ 1000 cps / ml).

  14. Patients with positive hepatitis C (HCV) antibody are not eligible for the study only if polymerase chain reaction shows negative HCVRNA.

  15. Clinically meaningful basic medicine, disease (e. g., dyspnea, pneumonia, pancreatitis, poorly controlled, poorly controlled diabetes, infection active or poorly controlled, or drug or alcohol abuse).

  16. Presence of severe neurological or psychiatric disorders, including dementia and epileptic seizures.

  17. He had an NCI-CTCAE grade 2 peripheral neuropathy. 18. Female patients during pregnancy or lactation. 19. Chronic bowel disease or short bowel syndrome. 20. Dihydropyrimidine dehydrogenase (DPD) enzyme deficiency. 21. Major cardiovascular diseases, such as New York Heart Association heart disease (grade II or higher), myocardial infarction within 3 months before randomization, unstable arrhythmia, or unstable angina pectoris.

  22. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction <50% must have an optimized stable medical regimen as determined by the treating physician, consulting a cardiologist if required.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 238 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival (3-y DFS) | 3-year
  The survival rate of patients without disease recurrence or death due to the disease progression patients at 36 months.

SECONDARY OUTCOMES:
Pathological complete response rate | Up to 6 months
  The proportion of patients with no tumor cells in the postoperative specimens
Overall Survival | Up to 5 years
  Time from the date of randomization until the date of death from any cause.
Objective Response Rate | Up to 6 months
  The rate of participants that achieve either a complete response (CR) or a partial response (PR).
Clinical complete response rate | Up to 36 months
  The disappearance of all detectable clinical and imaging evidence of a tumor after treatment
Incidence of adverse events | Up to 36 months
  Number of patients with AE, treatment-related AE (TRAE), immune-related AE (irAE), AE of special interest (AESI), serious adverse event (SAE) assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: WA He, Doctor, Principal Investigator — Shenzhen Peolple's Hospital

IPD SHARING:
Plan to Share IPD: No